CLINICAL TRIAL: NCT06046391
Title: A 12 Weeks,Multi-center,Randomized,Double-blind,Placebo-controlled Phase II Study to Evaluate the Efficacy and Safety of LP-003 in Adult Patients With Inadequately Controlled Moderate to Severe Seasonal Allergic Rhinitis Despite the Current Recommended Therapies
Brief Title: Efficacy and Safety of LP-003 in Moderate-to-severe Seasonal Allergic Rhinitis Adult
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Longbio Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P10-LP003-02
Record Dates: First submitted 2023-06-27; First posted 2023-09-21 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LP-003 dose 1 (Experimental): Eligible patients randomized to this arm received LP-003 subcutaneously for 8 weeks
  Interventions: Biological: LP-003 dose 1
- LP-003 dose 2 (Experimental): Eligible patients randomized to this arm received LP-003 subcutaneously for 8 weeks
  Interventions: Biological: LP-003 dose 2
- Placebo (Placebo Comparator): Eligible patients randomized to this arm received placebo subcutaneously for 8 weeks
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: LP-003 dose 1 — Liquid in vial
  Arms: LP-003 dose 1
Biological: LP-003 dose 2 — Liquid in vial
  Arms: LP-003 dose 2
Biological: Placebo — Liquid in vial
  Arms: Placebo

SUMMARY:
Allergic rhinitis (AR) affects large population worldwide, the most commonly used medication include anti-histamine, nasal spray and anti-LTRAs inhibitors (leukotriene receptor antagonists), Even after those first-line treatment, there is still a large number of patient (~20%) are not well/adequately controlled. Anti-IgE antibody has been approved to treat moderate to severe AR by PMDA/Japan in 2020, demonstrating the efficacy of IgE blockade in the treatment of allergic rhinitis. The current study presents a novel anti-IgE antibody (LP-003) with higher affinity to IgE, stronger efficacy and longer half-life.

DETAILED DESCRIPTION:
The purpose of this study was to evaluate the efficacy and safety of LP-003 in combination with SoC (nasal corticosteroids and/or anti-histamine) in adult patients with Moderate to Severe Seasonal Allergic Rhinitis, whose symptoms were inadequately controlled despite the current recommended therapies (nasal corticosteroids and/or anti-histamine) in the previous 2 pollen seasons.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 65 years at the screening period
2. Patients who met the diagnostic criteria of allergic rhinitis in Chinese Guidelines for the Diagnosis and Treatment of Allergic Rhinitis (revised edition, 2022) : a. Clinical symptoms: more than 2 (including 2 items) symptoms of sneezing, rhinorrhea, nasal congestion, nasal itching and other symptoms appear, which last or accumulate for more than 1h per day and may be accompanied by ocular symptoms such as itchy eyes/ tearing/ redness and burning heat sensation; b. Physical signs: pale, edema of the nasal mucosa and nasal watery discharge; c. Allergen detection: positive of at least 1 allergen skin prick test(SPT) and/or serum-specific IgE within 1 year before enrollment, or nasal provocation test positive
3. Had inadequately controlled symptoms (≥TNSS score of 6 and ≥ nasal congestion score of 2) of seasonal allergic rhinitis in last two years despite the use of nasal corticosteroid or in combination of one anti-histamine recommended by Guidelines.
4. Having any nasal symptom last for at least 2 days or any nasal and eye symptom last for at least one day, and ≥TNSS score of 1
5. Subjects (including partners) have no pregnancy and sperm, egg donation plan and voluntarily take one or more non-pharmaceutical measures for contraception, such as complete abstinence, intrauterine ring, partner ligation at period from drug administration to 6 months after the last study drug administration
6. voluntary participation in this trial and signing the informed consent form

Exclusion Criteria:

1. History of hypersensitivity to any content of the study drugs or its excipients..
2. Subjects with non-allergic rhinitis combined, such as drug rhinitis, vasomotor rhinitis, Nonallergic rhinitis with eosinophilia syndrome, acute and chronic sinusitis, rhinitis sicca anterior, atrophic rhinitis, obvious deviation of nasal septum
3. Subjects with perennial allergic rhinitis ( except for seasonal allergic rhinitis combined with perennial allergic rhinitis, which get attacks seasonally )
4. Subjects who have undergone nasal surgery or sinus surgery within 1 year before screening
5. Subjects who suffer from glaucoma, cataracts, herpes simplex keratitis, infectious conjunctivitis or currently and other eye infections ( Except for allergic conjunctivitis )
6. Subjects with active facial or systemic fungal, bacterial, viral or parasitic infection, and oral candida infection, who still require ongoing treatment
7. With clinically significant uncontrolled systemic disease (unstable ischemic heart disease, NYHA class III/IV left ventricular failure, arrhythmias, uncontrolled hypertension, cerebrovascular disease, neurodegenerative disease, other neurological disorders, uncontrolled hypothyroidism or hyperthyroidism and other autoimmune disorders, hypokalemia, hyperadrenergic status, diagnosed as a malignancy in the past, except for basal cell carcinoma or squamous cell skin cancer ) ; History of myocardial infarction (MI) within 1 year prior to the screening
8. In screening period: a) WBC < 2.5×10^9/L, b)AST or ALT > 2.0×ULN or TBIL > 1.5×ULN, c) Cr > 1.5×ULN
9. Subjects who have been treated by Omalizumab or other similar drugs within 6 months prior to the screening
10. Subjects who have taken systemic glucocorticoids within 4 weeks prior to the screening
11. Subjects who have taken intranasal glucocorticoids, mast cell membrane stabilizers, tricyclic antidepressants, leukotriene receptor antagonists, antihistamines within 1 week prior to the screening
12. Subjects who have taken traditional Chinese medicine for allergic rhinitis within 7 days prior to the screening
13. Subjects who have received allergen immunotherapy within half of year prior to the screening (in treatment), or who have received allergen immunotherapy within 3 years prior to the screening ( completed treatment )
14. During the study period, in addition to standard treatment concomitant drugs and salvage therapy drugs specified in the protocol. Subjects are prohibited from taking medications such as anticholinergics (oral and intranasal anticholinergics, including ipratropium nasal sprays), glucocorticoids, leukotriene receptor antagonists, antihistamines, mast cell membrane stabilizers, decongestants, nasal saline flushing, tricyclic antidepressants, antiallergic Chinese herbal medicines, immunosuppressants, immunomodulators and immunotherapy
15. Subjects with serious organic diseases such as heart, lung, liver, kidney
16. Subjects with poor compliance, such as poor medication compliance, inability to fill in diary cards correctly, and use of prohibited medications
17. Who combined with nerve and mental illness that could not or unwilling to follow the study, and with disabilities as prescribed by law (blind, deaf, mute, mentally disabled, mentally disabled, etc.)
18. Who plan to travel to other regions in which there is no allergic pollen during the study period for more than two consecutive days or three accumulated days
19. Pregnant or lactating women and women who plan pregnancy
20. Participated in other clinical studies within 3 months prior to the start of the study
21. Any condition that the investigator or primary physician believes may not be appropriate for participating the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2023-07-06 (Actual); Primary Completion 2023-10-19 (Actual); Study Completion 2024-08-06 (Actual)

PRIMARY OUTCOMES:
Mean nasal symptom score | peak pollen period(estimated average 4 weeks)
  Nasal symptoms (itchy, sneezing, rhinorrhea and nasal congestion) were recorded by the patient everyday in their e-Diary, on a scale of 0 (none) to 3 (intense/severe). Nasal symptom score (0-12 point) consisted of score for severity of itchy (0-3 point), sneezing (0-3 point), rhinorrhea (0-3 point) and nasal congestion (0-3 point).
  Peak pollen period was defined as the period between the first and last three consecutive days with ≥300 total pollen/1000 mm2 each day.

SECONDARY OUTCOMES:
Daily nasal symptom medication score | peak pollen period(estimated average 4 weeks)
  The daily nasal symptom medication score consisted of the sum of the daily nasal symptom severity score (0-12 points) and the daily nasal rescue medication score.
Daily nasal symptom medication score | pollen period(estimated average 10 weeks)
  The daily nasal symptom medication score consisted of the sum of the daily nasal symptom severity score (0-12 points) and the daily nasal rescue medication score.
  Pollen period was defined as the period between the first day when the total daily pollen count was ≥80 total pollen/1000 mm2 to the first day when the total daily pollen count was <80 total pollen/1000 mm2
Daily ocular symptom medication score | pollen period(estimated average 10 weeks)
  Ocular symptoms (itchy eyes/foreign body sensation/redness, tearing) were recorded by the patient everyday in their e-Diary, on a scale of 0 (none) to 3 (intense/severe). Ocular symptom score (0-6 point) consisted of score for severity of itchy eyes/foreign body sensation/redness (0-3 point) and tearing (0-3 point).
  The daily ocular symptom medication score consisted of the sum of the daily ocular symptom severity score (0-6 points) and the daily ocular rescue medication score.

CONTACTS AND LOCATIONS:
Locations (17):
- China (17):
  - Beijing Shijitan Hospital, Beijing, Beijing Municipality
  - Dongfang Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Zhengzhou central hospital, Zhengzhou, Henan
  - Changchun University of Chinese Medicine Affiliated Hospital, Changchun, Jilin
  - Tonghua central hospital, Tonghua, Jilin
  - Yan Bian Chao Yi Hospital, Yanbian, Jilin
  - Yanbian University hospital, Yanji, Jilin
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Yinchuan Peoples Hospital, Yinchuan, Ningxia
  - Zibo central hospital, Zibo, Shandong
  - Linfen Peoples Hospital, Linfen, Shanxi
  - Second hospital of Shanxi Medical University University, Taiyuan, Shanxi
  - The First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Xidian group hospital, Xi’an, Shanxi
  - Tianjin Peoples Hospital, Tianjing, Tianjing

IPD SHARING:
Plan to Share IPD: No